CLINICAL TRIAL: NCT00763464
Title: Coronary Artery Disease in Postmenopausal Women. Comparison of Myocardial Szintigraphy With Sress-Echocardiography and Stress-MRI.
Brief Title: Coronary Artery Disease (CAD) in Postmenopausal Women
Acronym: FEMCAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Michael Becker, MD, Medical Clinic I, Medical Faculty of the RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAD female 2006-MB
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Postmenopausal Women; Stable Angina Pectoris
Keywords: Coronary Artery Disease; ischemia diagnostic
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: stress-echocardiography — stress-echocardiography will be performed once using Adenosin (140 µg/kg/min over 6 Minutes) and a contrast agent (SonoVue)
Procedure: stress-MRI — stress-MRI will be performed once using Adenosin (140 µg/kg/min over 6 Minutes)and a contrast agent (Gadovist)

SUMMARY:
Aim of this study is the determination of a valid procedure for ischemia diagnositc in postmenopausal women.

DETAILED DESCRIPTION:
In order to investigate which ischemia diagnostic presents which sensitivity and specificity for postmenopausal women, 100 consecutive patients presenting to our abmulance with stable angina pectoris and indication for myocardial szintigraphy will be enrolled in this study. An addidional stress-echocardiography and stress-MRI will be performed in this patients before they will reiceve their again routine coronay angiography.

The different methods for ischemia diagnostic will be compared in order to determine the most valid method for this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women presenting to the hospital with stable Angina pectoris complaints and an indication for myocardial szintigraphy

Exclusion Criteria:

* CABG
* Pacemaker or other metal implants
* Chronic bronchitis
* Asthma bronchiale
* Arterial Hypotension

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
comparision of different ischemia diagnostic methods | before routine coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, MD, Principal Investigator — Medical Faculty of the RWTH Aachen University
Locations (1):
- Department of Cardiology, RWTH Aachen University Hospital, Aachen, Germany